CLINICAL TRIAL: NCT05198349
Title: First-in-Human Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Activity of M1069 in Participants With Metastatic or Locally Advanced Unresectable Solid Tumors
Brief Title: First in Human Study of M1069 in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Overarching portfolio-level review of the company's oncology pipeline resulted in early termination of the study. The study was not terminated due to safety.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS201929_0032
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Metastatic or Locally Advanced Unresectable Solid Tumors
Keywords: Adenosine antagonist; Adenosine receptor A2A/A2B antagonist; M1069
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- M1069 (Experimental)
  Interventions: Drug: M1069

INTERVENTIONS:
Drug: M1069 — Participants received escalated oral dose of M1069, twice daily (BID) until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from study intervention.

SUMMARY:
The main purpose of this study was to determine the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and early signs of efficacy of M1069 in participants with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had histologically or cytologically proven locally advanced or metastatic solid malignancies and who are refractory to or have progressed under standard treatment or for whom standard treatment is not expected to deliver clinical benefit
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at Screening
* Adequate hematological function, hepatic function and renal function
* Ability to swallow oral dose forms (for example [e.g.] capsules)
* Fresh tumor biopsies mandatory for participants at Dose level 2 (DL2) and 6 participants upon potential determination of Recommended Dose for Expansion (RDE). Providing consent to fresh tumor biopsies taken during the Screening period and an on-treatment biopsy is mandatory
* Life expectancy of at least 12 weeks according to Investigator judgement
* Measurable disease according to The Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Persisting toxicity related to prior therapy Grade greater than (>) 1 National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0, however, alopecia, sensory neuropathy hypothyroidism and diabetes mellitus Grade less than or equal to (<=) 2, despite treatment, are allowed
* Prior organ transplantation including allogeneic stem cell transplantation
* Participants with known brain metastases, except those meeting the following criteria: a) Brain metastases that have been treated locally and are clinically stable for at least 4 weeks prior to the start of treatment; b) No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
* Participants must be either off steroids or on a stable or decreasing dose of < 10 milligrams (mg) daily prednisone (or equivalent)
* Current significant cardiac conduction abnormalities, including corrected QT interval (QTcF, corrected with Fridericia formula) prolongation of > 470 milliseconds (ms) or impaired cardiovascular function, ventricular tachycardia (including Torsades de Pointes), or a history of paroxysmal atrial fibrillation, serious cardiac arrhythmia and family history of sudden death or long QT syndrome
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent including but not limited to inflammatory bowel diseases, autoimmune hepatitis, interstitial lung disease of immunologic origin, systemic lupus erythematosus, et cetera (etc.), with the following exceptions: a) Participants with diabetes type I, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
* Significant acute or chronic fungal, bacterial and/or viral infections requiring systemic therapy including coronavirus disease of 2019 (COVID-19)
* Known hypersensitivity to the trial treatment or to one or more of the excipients
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Safety Profile as Assessed by Incidence of Adverse Events (AEs), Treatment-Related AEs and Dose-Limiting Toxicities (DLTs) | Time from first dose of study drug up to planned assessment at 18.2 months

SECONDARY OUTCOMES:
Pharmacodynamic Assessment by Phosphorylated cAMP Response Element-binding Protein (pCREB) Level in ex-vivo Stimulated Blood | Pre-dose up to 8 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 8; Pre-dose on Cycle 2 Day 1 (each cycle is of 21 days)
Change from Baseline in Tumor Microenvironment (TME) in Available Paired Tumor Biopsies at Cycle 2 Day 15 | Baseline, Cycle 2 Day 15 (each cycle is of 21 days)
Pharmacokinetic (PK) Plasma Concentrations of M1069 | Pre-dose up to 24 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 8 (each cycle is of 21 days)
Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), as Assessed by Investigator | Time from first dose of study drug up to planned assessment at 18.2 months
Duration of Response (DoR) | Time from first dose of study drug up to planned assessment at 18.2 months
Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), as Assessed by Investigator | Time from first dose of study drug up to planned assessment at 18.2 months
Change from Baseline in Corrected QT (QTc) Interval Over Time | Pre-dose (Baseline) up to 8 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 8 (each cycle is of 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (3):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Sarah Cannon Research Institute (SCRI) (The SCRI Oncology Research Consortium), Nashville, Tennessee
- Princess Margaret Cancer Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201929_0032
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html